CLINICAL TRIAL: NCT05648214
Title: A Three-Part, Phase 1, Randomized, Double-blind, Placebo-Controlled, Single and Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of ALN-PNP, an siRNA Targeting PNPLA3, in Healthy Adults and Adult Participants With MASLD
Brief Title: A Trial to Learn if ALN-PNP is Safe and Well Tolerated in Healthy Adults and Adult Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-PNP-HV-2227
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Keywords: Liver steatosis; Fibrosis; Hepatocytes; Non-Alcoholic Steatohepatitis (NASH); Non-Alcoholic Fatty Liver Disease (NAFLD); Metabolic dysfunction-Associated Steatohepatitis (MASH)
MeSH Terms: conditions — Fatty Liver; Fibrosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Part A: Sequential ascending dose Part B and Part C: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Cohorts (Experimental)
  Interventions: Drug: ALN-PNP; Drug: Placebo (PB)
- Part A: Optional Cohort (Experimental)
  Interventions: Drug: ALN-PNP; Drug: Placebo (PB)
- Part A: JPN Cohorts (Experimental)
  Interventions: Drug: ALN-PNP; Drug: Placebo (PB)
- Part B: Cohorts (Experimental)
  Interventions: Drug: ALN-PNP; Drug: Placebo (PB)
- Part C: Cohorts (Experimental)
  Interventions: Drug: ALN-PNP; Drug: Placebo (PB)

INTERVENTIONS:
Drug: ALN-PNP — Administered per the protocol
Drug: Placebo (PB) — Administered per the protocol

SUMMARY:
This study is researching an experimental drug called ALN-PNP (called "study drug"). This is a first in human study. The study drug is not approved by any public health agency such as the United States Food and Drug Administration (FDA) for any kind of treatment.

This study consists of 3 parts. Part A is focused on healthy participants. Parts B and C of the study are focused on participants who are known to have MASLD and a specific variant of the PNPLA3 gene.

The aim of the study is to see how safe, tolerable and effective the study drug is.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug (Parts A, B and C)
* How much study drug (Parts A, B and C) and study drug metabolites (byproduct of the body breaking down the study drug) (Parts B and C) are in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects) (Part A, B and C)
* Explore impact of Japanese ethnicity on safety and PK (Pharmacokinetics, or study of what the body does to the drug) of single doses of ALN-PNP over time (Part A)
* How the study drug works to change liver fat content in MASLD (Part B and C)
* Better understanding of the study drug and MASLD (Part B and C)

ELIGIBILITY:
Key Inclusion Criteria:

Part A (Healthy Adults):

1. From 18 to 55 years of age
2. For Japanese cohorts ONLY; the Japanese participant must:

   1. Be Japanese, born in Japan, and have both biologic parents and 4 biologic grandparents who are ethnically Japanese and born in Japan
   2. Have maintained a Japanese lifestyle, with no significant change since leaving Japan, including having access to Japanese food and adhering to a Japanese diet
   3. Be living <10 years outside of Japan
3. Has a body mass index between 18 and 32 kg/m^2, inclusive, at the screening visit
4. Is judged by the investigator to be in good health, as described in the protocol
5. Is in good health based on laboratory safety testing obtained at the screening visit and approximately within 24 hours prior to administration of study drug

Part B and Part C (Participants with MASLD):

1. Part B: From 18 to 65 years of age
2. Part C: From 18 to 75 years of age
3. Body mass index (BMI) from 23.0 kg/m2 to 40.0 kg/m2, inclusive, for East Asians (including but not limited to South Koreans, Chinese, Taiwanese, and Japanese) and BMI from 27.0 kg/m2 to 40.0 kg/m2, inclusive, for any other ethnicity at screening visit 1
4. Liver fat content ≥8.5% as measured by MRI-PDFF at screening visit 3

Key Exclusion Criteria:

Part A:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, neurological, or dermatologic disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation
2. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Hospitalized for any reason within 30 days of the screening visit
4. Using the Modification of Diet in Renal Disease equation, has a glomerular filtration rate as described in the protocol at the screening visit
5. Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin above the upper limit of normal (ULN) range
6. Is a current smoker or former smoker, including e-cigarettes, who stopped smoking within 3 months prior to the screening visit
7. Has a history of alcohol or drug abuse per investigator opinion
8. Is positive for hepatitis C antibody and if so, positive for qualitative (ie, detected or not detected) hepatitis C virus ribonucleic acid (RNA) test at the screening visit

Part B and Part C:

1. Evidence of other forms of known chronic liver disease, as defined in the protocol
2. Has a contraindication to MRI examinations, as defined in the protocol
3. History of Type 1 diabetes
4. Has lost or gained more than 4.0% body weight over the 3 months prior to or during the screening period
5. Has known human immunodeficiency virus (HIV) infection, evidence of current or chronic hepatitis B virus (HBV) infection, or current or chronic hepatitis C virus (HCV) infection, as defined in the protocol
6. Bariatric surgery within approximately 5 years (Part B) or 3 years (Part C) prior or planned during the study period

NOTE: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to Day 253
Severity of TEAEs | Up to Day 253

SECONDARY OUTCOMES:
Concentration of ALN-PNP and potential major metabolite(s) in plasma | Up to Day 253
Incidence of Anti-Drug Antibodies (ADAs) to ALN-PNP | Up to Day 253
Magnitude of ADAs to ALN-PNP | Up to Day 253
Change in Low-Density Lipoprotein (LDL) | Baseline up to Day 169
  Part A
Change in High-Density Lipoprotein (HDL) | Baseline up to Day 169
  Part A
Change in TriGlyceride (TG) | Baseline up to Day 253
Change in Apolipoprotein B (ApoB) | Baseline up to Day 253
Change in liver fat fraction by Magnetic Resonance Imaging derived Proton-Density Fat Fraction (MRI-PDFF) | Baseline up to Day 253
  Part B and Part C
Change in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline up to Day 253
  Part B and Part C
Change in High-Density Lipoprotein Cholesterol (HDL-C) | Baseline up to Day 253
  Part B and Part C
Change in Lipoprotein (a) (Lp[a]) | Baseline up to Day 253
  Part B and Part C
Change in Apolipoprotein A1 (ApoA1) | Baseline up to Day 253
  Part B and Part C
Change in small dense Low-Density Lipoprotein (sdLDL) | Baseline up to Day 253
  Part C

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- United States (6):
  - California Clinical Trials Medical Group, Glendale, California
  - Velocity Clinical research, Los Angeles, California
  - Genoma Research Group, Inc, Miami, Florida
  - Med Research of Florida, LLC, Miami, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Pioneer Research Solutions, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/